CLINICAL TRIAL: NCT06166069
Title: Early Surgical Outcomes in the Use of Hybrid Mesh for Incisional Hernia Repair: Results From a Multicenter Italian Study
Acronym: SHIELD
Status: Completed | Type: Observational
Sponsor: Azienda Sanitaria Locale Napoli 2 Nord (Other)
Responsible Party: Principal Investigator, Francesco Pizza, PhD, Md, Azienda Sanitaria Locale Napoli 2 Nord
Other Study IDs: 202318
Record Dates: First submitted 2023-12-01; First posted 2023-12-12 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Hernia; Incisional Hernia; Laparoscopic
Keywords: Hernia
MeSH Terms: conditions — Hernia; Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: Intraperitoneal Onlay Mesh(IPOM) Plus (GroupA) the laparoscopic closure of the hernia defect will be then performed with detached stitches, non-resorbable 1/0 suture with running intracorporeal suture or intra/extracorporeal interrupted suture
- B: Intraperitoneal Onlay Mesh(IPOM) standard (Group B) no defect closure will be performed.

SUMMARY:
Background: Ventral hernia repair poses challenges for surgeons due to controversies in approach, patient selection, and mesh selection. The GORE® SYNECOR Intraperitoneal (IP) Biomaterial, a hybrid mesh, aims to balance durability and infection risk.

Objective: To analyze extended-term outcomes of using the Intaperitoneal device for ventral and incisional hernia repair.

Methods: Retrospective analysis of patients undergoing surgery in eight Italian Surgery Centers, evaluating pIPOM and sIPOM techniques with GORE® SYNECOR IP Biomaterial. Preoperative evaluations included anthropometric measurements, comorbidities, CT scans, and GIQLI assessments. Surgical procedures and interventions were recorded. Postoperative complications, GIQLI changes, cosmesis, hernia recurrence, and mesh bulging were assessed.

DETAILED DESCRIPTION:
The management of ventral hernias, whether they are primary or incisional, presents a significant challenge for abdominal wall surgeons. Laparoscopic ventral hernia repair has become a widely accepted technique on a global scale, with literature reporting favorable outcomes, even over the long term. Nevertheless, various substantial controversies have emerged concerning the ideal approach and patient selection and "ideal mesh". Permanent mesh materials with a macro-porous structure have demonstrated excellent durability, a low risk of infection in ventral hernia repair. Nevertheless, hernia recurrences and complications can still occur. The use of absorbable mesh materials may reduce the risk of infectious complications and the need for mesh removal. However, it might be associated with a higher likelihood of long-term recurrence when compared to permanent materials.

In response to these challenges, hybrid mesh materials, combining both absorbable and permanent components, have been developed to strike a balance between achieving long-term durability and minimizing the risk of infection or "Mesh removal". These hybrid meshes can be utilized either intraperitoneally or extra-peritoneally depending on their composition.

One example of such a hybrid mesh is the GORE® SYNECOR Intraperitoneal Biomaterial (referred to as the device), manufactured by W.L. Gore & Associates, Inc. in Flagstaff, AZ. This composite mesh comprises a bioabsorbable 3D web scaffold and a permanent dense polytetrafluoroethylene (PTFE) monofilament macro-porous knit. The device is specifically designed for intraperitoneal placement, using either an underlay or intraperitoneal onlay technique.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* Clean wounds
* Informed consent
* Patients affected by Incisional and Ventral Hernia
* Elective surgery
* Hernia size between 3 e 10 cm

Exclusion Criteria:

* age < 18 years;
* Life expectancy < 24 months (as estimated by the operating surgeon), -
* Pregnancy
* Immunosuppressant therapy within 2 weeks before surgery
* Clean-contaminated and contaminated, dirty wounds
* Cirrhosis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Enrolled participants were allocated to either the pIPOM or sIPOM Groups based on the routine surgical practices of each center. In Group A, (IH) repairs were performed with the closure of the fascia using sutures (pIPOM). In Group B, laparoscopic IH repairs were carried out without closing the fascia (sIPOM). The choice of prosthesis dimensions was customized, with a minimum requirement of at least a 5 cm overlap.
  Postoperative complications, including morbidity (assessed according to the Clavien-Dindo classification [9]), mortality, length of hospital stay, and surgical reinterventions, were documented. All patients underwent regular follow-up at 1, 3, 6, and 12 months. During these follow-up visits, anthropometric measurements were conducted.
Sampling Method: Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-11-18 (Actual)

PRIMARY OUTCOMES:
Number of patients affected by Superficial surgical site infections | Within 30 days postoperatively
  Superficial infections according to Clavien-Dindo criteria
Number of patients affected by Deep surgical site infections | Within 30 days postoperatively
  Deep surgical site infections according to Clavien-Dindo criteria
Number of patients affected by organ space infections | Within 30 days postoperatively
  Organ space infections according to Clavien-Dindo criteria
Number of patients affected by Surgical Site Occurence | Within 30 days postoperatively
  Surgical Site Occurence Reported according to the Ventral Hernia Working Group (VHWG) definitions
Postoperative pain | Postoperative pain will be recorded according to visual analogue scale Visual Analogue Scale at 1 month.
  Postoperative pain will be recorded according to the Visual Analogue Scale (VAS). The Visual Analogue Scale (VAS) measures pain intensity. The Visual Analogue Scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Postoperative pain | Postoperative pain will be recorded according to visual analogue scale Visual Analogue Scale at 6 month.
  Postoperative pain will be recorded according to the Visual Analogue Scale (VAS). The Visual Analogue Scale (VAS) measures pain intensity. The Visual Analogue Scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Postoperative pain | Postoperative pain will be recorded according to visual analogue scale Visual Analogue Scale at 12 month.
  Postoperative pain will be recorded according to the Visual Analogue Scale (VAS). The Visual Analogue Scale (VAS) measures pain intensity. The Visual Analogue Scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

SECONDARY OUTCOMES:
Rate of Incisional Hernia at Clinical examination | Patients are postoperatively examined at 1 months.
  Clinical examination: Incisional Hernia is clinically defined as any visible or palpable ''blowout'' in site of incisional hernia treated
Rate of Incisional Hernia at Clinical examination | Patients are postoperatively examined at 6 months.
  Clinical examination: Incisional Hernia is clinically defined as any visible or palpable ''blowout'' in site of incisional hernia treated
Rate of Incisional Hernia at Clinical examination | Patients are postoperatively examined at 12 months.
  Clinical examination: Incisional Hernia is clinically defined as any visible or palpable ''blowout'' in site of incisional hernia treated
Rate of Incisional Hernia at ultrasonographic examination | Patients are postoperatively examined at 1 months.
  An abdominal ultrasonography with the patient lying prone, will be performed in in all patients (symptomatic or asymptomatic) providing any valuable information about Hernia Recurrence onset. Valsalva maneuver will be performed during the ultrasonography scan. Size and location of all imaging detected Hernia Recurrence will be recorded, as well as any other patient's complaint.
Rate of Incisional Hernia at ultrasonographic examination | Patients are postoperatively examined at 6 months.
  An abdominal ultrasonography with the patient lying prone, will be performed in in all patients (symptomatic or asymptomatic) providing any valuable information about Hernia Recurrence onset. Valsalva maneuver will be performed during the ultrasonography scan. Size and location of all imaging detected Hernia Recurrence will be recorded, as well as any other patient's complaint.
Rate of Incisional Hernia at ultrasonographic examination | Patients are postoperatively examined at 12 months.
  An abdominal ultrasonography with the patient lying prone, will be performed in in all patients (symptomatic or asymptomatic) providing any valuable information about Hernia Recurrence onset. Valsalva maneuver will be performed during the ultrasonography scan. Size and location of all imaging detected Hernia Recurrence will be recorded, as well as any other patient's complaint.

CONTACTS AND LOCATIONS:
Locations (1):
- francesco Pizza, Naples, Italy

REFERENCES:
- [Derived] Pizza F, Iuppa A, Maida P, Pilone V, Crucitti A, Carmen TPM, Morini L, Marin JN, Petitti T, Bertoglio C, Marte G, Sordelli I, Gili S, Lucido FS, Busciano L, D'Antonio D, Docimo L, Gambardella C. Postoperative outcomes and wound events in incisional hernia repair using hybrid mesh: results from a prospective multicenter italian study. Hernia. 2025 Feb 18;29(1):94. doi: 10.1007/s10029-025-03285-z. PMID 39966208